CLINICAL TRIAL: NCT01923974
Title: The Analgesic Effects of Melatonin: A Randomized, Placebo-controlled, Double-blinded Study on Healthy Volunteers
Brief Title: The Analgesic Effects of Melatonin
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Lars Peter Holst Andersen (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Sponsor-Investigator, Lars Peter Holst Andersen, Ph.d. fellow, Herlev Hospital
Organization: Herlev Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: CPO-2013
Record Dates: First submitted 2013-08-08; First posted 2013-08-16 (Estimated); Last update posted 2014-10-22 (Estimated); Status verified 2014-10

CONDITIONS: Analgesia; Antihyperalgesia
MeSH Terms: conditions — Agnosia | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): IV formulation
  Interventions: Drug: Placebo
- Melatonin 10 mg (Active Comparator): IV formulation, Melatonin 10 mg
  Interventions: Drug: Melatonin 10 mg
- Melatonin 100 mg (Active Comparator): IV formulation, Melatonin 100 mg
  Interventions: Drug: Melatonin 100 mg

INTERVENTIONS:
Drug: Melatonin 10 mg
  Arms: Melatonin 10 mg
Drug: Melatonin 100 mg
  Arms: Melatonin 100 mg
Drug: Placebo
  Arms: Placebo

SUMMARY:
A study investigating the analgesic effect of melatonin in a human heat injury model using quantitative sensory testing.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males aged between 20 and 40 years

Exclusion Criteria:

* Under aged/minors
* Does not speak or understand danish
* Alcohol or abuse of medicines
* Prior QST-trial within the last 2 month
* Prior medical trail within the last month
* Serious comorbidity (ASA-class 3-4)
* Chronic pain (defined by analgesic treatment) Shift-work or night work within the last 14 days Known sleep-disorder

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2013-08; Primary Completion 2014-06 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Pain (VAS) | During burn injury. 1 hours following melatonin/placebo administration
Change in areas of secondary hyperalgesia | 1,2,4,6 hours following burn injury, which corresponds to 2,3,5 and 7 hours after melatonin/placebo-administration
  Areas of secondary hyperalgesia will be assessed by quantitative sensory testing

SECONDARY OUTCOMES:
Change in erythema/oedema assessed by ultrasound | 1,2,4,6 hours following burn injury, which corresponds to 2,3,5 and 7 hours after melatonin/placebo-administration
Thermal thresholds assessed by quantitative sensory testing | 1,2,4,6 hours following burn injury, which corresponds to 2,3,5 and 7 hours after melatonin/placebo-administration
Mechanical thresholds assessed quantitative sensory testing | 1,2,4,6 hours following burn injury, which corresponds to 2,3,5 and 7 hours after melatonin/placebo-administration

CONTACTS AND LOCATIONS:
Overall Officials: Lars P.H. Andersen, MD, Principal Investigator — Herlev Hospital
Locations (1):
- Multidisciplinary Pain Center 7612, Neuroscience Center, Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Derived] Andersen LP, Werner MU, Rosenkilde MM, Harpsoe NG, Fuglsang H, Rosenberg J, Gogenur I. Pharmacokinetics of oral and intravenous melatonin in healthy volunteers. BMC Pharmacol Toxicol. 2016 Feb 19;17:8. doi: 10.1186/s40360-016-0052-2. PMID 26893170